CLINICAL TRIAL: NCT04290845
Title: Relief-Hybrid: A Behavioral Intervention for Depression and Chronic Pain in Primary Care
Brief Title: A Behavioral Intervention for Depression and Chronic Pain in Primary Care (Relief-Hybrid)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated due to COVID-19. No study participants were enrolled.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-10020967; 5P50MH113838 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Depression
Keywords: Chronic Pain; Depression; Primary Care; Older Adults; Middle Aged
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants will be blinded as to who is receiving Relief-Hybrid and who is receiving Usual Care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relief-Hybrid (Experimental): Relief-Hybrid relies on a neurobiological model to simplify its behavioral targets and uses mobile technology to augment its interventions. Relief was co-developed with our primary care partners with the goal to be usable by non-physician clinicians of primary care offices eligible to provide billable services.
  Interventions: Behavioral: Relief-Hybrid
- Referral to Mental Health/Usual Care (No Intervention): Continuation of medical attention and treatment provided by physicians and other medical professionals at the primary care practice. Referral for mental health based on clinical indication. Participants receive an educational booklet on pain.

INTERVENTIONS:
Behavioral: Relief-Hybrid — A 9-week behavioral intervention for primary care patients designed to reduce depression and pain-related disability.
  Arms: Relief-Hybrid

SUMMARY:
Chronic pain and depression frequently co-exist in late and mid-life and contribute to increased disability, high health care costs, psychiatric comorbidity, and suicide. Older and middle-aged depressed-pain patients: a) are mainly treated in primary care practices; and b) are often prescribed medication, which increases the risk for addiction to opioids and benzodiazepines. Despite the need and desire by the patients and providers for primary care behavioral intervention, behavioral interventions are scarce in primary care.

To address this need, Relief-Hybrid was created. Subjects are randomized to either the Relief-Hybrid intervention or to Referral to Mental Health/Usual Care. Subjects in both arms will complete research assessments at 6, 9, and 12 weeks. Subjects in the Relief-Hybrid arm will receive 5 weekly sessions with the study therapist (licensed social workers, LCSWs) and 4 self-administered, mobile technology-assisted sessions.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* PHQ-9 score greater or equal to 10
* Chronic pain (non-cancer related, most days over the past 3 months)
* Capacity to consent

Exclusion Criteria:

* DSM-5 Axis 1 diagnoses other than depression and anxiety disorders
* Montreal Cognitive Assessment (MoCA) < 24
* Active suicidal ideation (MADRS item #10 greater or equal to 4
* Severe or life-threatening medical illness
* Patients on psychotropics, opioids or benzodiazepines will be included if they do not meet DSM-5 criteria for opioid, anxiolytics or other substance abuse disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms, as measured by the Montgomery Asberg Depression Rating Scale (MADRS) | Baseline, 6, 9, and 12 weeks
  The MADRS is a 10 item questionnaire assessing severity of depression by scoring participants on mood, anxiety, sleep, concentration, appetite, and suicidal thoughts. The lowest score is 0, no depression symptoms, and the highest possible score is 60, severe depression symptoms.
Change in Pain-Related Disability, as measured by the Roland-Morris Disability Questionnaire (RMDQ) | Baseline, 6, 9, and 12 weeks
  The RMDQ includes a scale assessing how much pain the participant has experienced in the past week, with 0 meaning no pain and 10 meaning pain as bad as he/she can imagine.
  The RMDQ also includes a series of questions related to pain disability, with 0 indicating no pain-related disability, and 24 indicating severe pain-related disability.
Change in Mood, as measured by the Daily Photographic Affect Meter (PAM) | Daily for 12 Weeks
  The PAM is used for assessing mood and emotional state. Participants can either score a "positive" or "negative" affect value.

SECONDARY OUTCOMES:
Interoceptive Awareness, as measured by the Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline, 6, 9, and 12 weeks
  This assessment contains 32 questions measuring 8 areas of manifestations of emotions, including noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. The scores for the questions associated with each of the 8 domains are averaged, with a score of 0 indicating "Never" and a score of 5 indicating "Always"
Affect, as measured by the Positive and Negative Affect Schedule (PANAS). | Baseline, 6, 9, and 12 weeks
  This scale consists of a series of 60 words and phrases and participants rate to what extent they have felt that way in the past week. The words are separated into 13 areas: general negative affect, fear, sadness, guilt, hostility, shyness, fatigue, general positive affect, joviality, self-assurance, attentiveness, serenity, and surprise. The scores range from 1 (very slightly/not at all), to 5 (extremely) for each word and each area is summed for the final score.
Mood, as measured by the Mood Likert Scale | Daily for 12 weeks
  This scale rates current sadness, ranging from 0 (not sad) to 10 (most sad). It also rates interest or pleasure in doing things, ranging from 0 (no interest or pleasure) to 10 (greatest interest or pleasure).
Pain, as measured by the Pain Likert Scale | Daily for 12 weeks
  This scale rates current pain, ranging from 0 (no pain) to 10 (worst pain possible).
Stress, as measured by the Stress Likert Scale | Daily for 12 weeks
  This scale rates current stress, ranging from 0 (no stress at all) to 10 (great stress).
Activities Monitoring | Daily for 12 Weeks
  Activities monitoring through a phone application; measuring distance covered daily by the participant during the week.
Activities Monitoring | Daily for 12 Weeks
  Activities monitoring through a phone application; measuring number of places visited daily during the week.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Weill Cornell Internal Medical Associates (WCIMA), New York, New York
  - Iris Cantor Men's and Women's Health Centers, New York, New York
  - Irving Sherwood Wright Center, New York, New York
  - Weill Cornell Institute of Geriatric Psychiatry, Weill Cornell Medicine, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: https://nda.nih.gov/